CLINICAL TRIAL: NCT06437275
Title: The Degree of Knowledge and Attitude of Egyptian Physicians Regarding Emergency Treatment of Traumatic Dental Injuries: Cross Sectional Study
Brief Title: The Degree of Knowledge and Attitude of Egyptian Physicians Regarding Emergency Treatment of Traumatic Dental Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nour Ziad Al-Tabbaa, Principal investigator - Dr. Nour Ziad Al-Tabbaa, Cairo University
Other Study IDs: knowloedge and attitude
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Dental Injuries
Keywords: Traumatic dental injuries; awareness; knowledge; attitude
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire for the degree of knowledge and attitude — Questionnaire for the degree of knowledge and attitude of Egyptian physicians regarding emergency treatment of traumatic dental injuries.

SUMMARY:
This study intends to evaluate physicians' fundamental knowledge and attitude regarding the management of TDIs in Egypt. A convenience sample of physicians will be enrolled in this cross-sectional study, and they will be asked to complete a validated questionnaire. The questionnaire includes demographic questions, two case scenarios involving crown fractures and the avulsion of permanent teeth, and self-evaluation questions.

DETAILED DESCRIPTION:
Several epidemiological studies continue to show significant levels of dental trauma in many countries. In industrialized countries, about one in five children experience a traumatic dental injury (TDI) to permanent teeth before leaving school.

Primary care providers (e.g., family physicians, pediatricians, emergency medicine physicians and nurses) can play an important role in offering primary care following dentofacial trauma, especially for rural populations with limited access to dentists.

Several global studies indicate that physicians and even pediatricians lacked the emergency management knowledge to deal with traumatic dental injuries (TDIs). Emphasizing the fact that medical students are not well educated or trained to manage TDIs.

To the best of our knowledge, no study has been conducted in Egypt to investigate physicians' knowledge and attitudes addressing traumatic dental injury.

ELIGIBILITY:
Inclusion Criteria:

Physicians who accept to participate.

Exclusion Criteria:

Physicians who refuse to participate.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are family medicine, pediatricians, emergency doctors and other specialties in Cairo and Ain Shams University in Egypt.
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The degree of knowledge and attitude of Egyptian physicians. | 2 months
  Evaluate Egyptian physicians knowledge and attitude regarding the management of dental trauma using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sherien Badr, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Al Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
evaluate physicians' fundamental knowledge and attitude regarding the management of TDIs in Egypt.

REFERENCES:
- [Result] Al-Haj Ali SN, Farah RI, Alhariqi S. Knowledge and Attitudes of Saudi Medical Students about Emergency Management of Traumatic Dental Injuries. Int J Environ Res Public Health. 2022 Oct 31;19(21):14249. doi: 10.3390/ijerph192114249. PMID 36361130
- [Result] Al Barkhati S, Al Mullahi A. Knowledge and Awareness of Emergency Medical Physicians on the Management of Traumatic Dental Avulsion at Sultan Qaboos University Hospital. Sultan Qaboos Univ Med J. 2023 Nov;23(4):479-484. doi: 10.18295/squmj.5.2023.030. Epub 2023 Nov 30. PMID 38090234
- [Result] Sari MBD, Sari E, Bal C, Aksoy M. Evaluation of the knowledge level of pediatricians on dental trauma and their awareness of the ToothSOS mobile application: A cross sectional study. Dent Traumatol. 2024 Apr;40(2):195-203. doi: 10.1111/edt.12895. Epub 2023 Oct 18. PMID 37849392
- [Result] Raoof M, Vakilian A, Kakoei S, Manochehrifar H, Mohammadalizadeh S. Should medical students be educated about dental trauma emergency management? A study of physicians and dentists in Kerman Province, Iran. J Dent Educ. 2013 Apr;77(4):494-501. PMID 23576595
- [Result] Iyer SS, Panigrahi A, Sharma S. Knowledge and Awareness of First Aid of Avulsed Tooth among Physicians and Nurses of Hospital Emergency Department. J Pharm Bioallied Sci. 2017 Apr-Jun;9(2):94-98. doi: 10.4103/jpbs.JPBS_343_16. PMID 28717331